CLINICAL TRIAL: NCT03203213
Title: Musitox® Project: Consumption of Psychoactive Substances at Music Festivals in Aquitaine
Acronym: Musitox®
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Regional Health Agency New Aquitaine (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHUBX 2017/12
Record Dates: First submitted 2017-06-27; First posted 2017-06-29 (Actual); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Poisoning by Psychoactive Substances
Keywords: Poisoning; Psychoactive substances
MeSH Terms: conditions — Poisoning | interventions — Urination

STUDY DESIGN:
Intervention Model Description: monocentric study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional arm (Experimental): * Sampling of a few additional drops of blood and sending this sample for analysis and identification of a possible toxic cause by psychoactive substance in relation to the clinical picture presented by the patient
  * Oriented hair removal is also carried out if possible (small wick cut and not torn the size of a pencil mine of paper taken at the level of the occipital region). This technique has been used many times, and evaluates the previous consumption (memory consumption)
  * A urine sample is taken if possible.
  Interventions: Procedure: Sampling of a few drops of blood, lock of hair and urine

INTERVENTIONS:
Procedure: Sampling of a few drops of blood, lock of hair and urine — Sampling of a few additional drops of blood to deposit them on blotting paper (DBS: Dried Blood Spot) ad hoc and to send this sample for analysis and identification of a possible toxic cause by psychoactive substance in relation to the clinical picture presented by the patient. An oriented capillary sampling is also performed if possible. Similarly a urine sample is taken if possible.

SUMMARY:
Poisoning by psychoactive substances is increasingly common in Europe and can be responsible for deaths. These substances, also called "festive drugs", circulate among other places in festive gatherings (night clubs, concerts, free music, feria, etc.). The main objective of this study is to determine the molecules that circulate in festive events in Aquitaine, in order to implement prevention actions by looking at whether the circulating substances vary with the style of event.

DETAILED DESCRIPTION:
Poisoning by psychoactive substances is increasingly common in Europe and can be responsible for deaths. These substances, also called "festive drugs", circulate among other places in festive gatherings (night clubs, concerts, free music, feria, etc.).

There is also a significant increase in the number of new psychoactive substances (NSPs) whose toxicity is unknown: by 2014, 101 new substances were detected for the first time in Europe. These molecules, because of this regular and rapid emergence, are not included in the narcotics list, in the great majority of cases.

Poison control centers, as well as addictovigilance centers, are regularly called upon for serious poisoning resulting in hospitalization, for which analytical evidence is most often missing or difficult to obtain. The lack of documentation, both analytical and clinical, of these files limits its expertise. As a result, medical knowledge, in particular clinical knowledge, progresses little which limits the efficiency of the management of these poisonings.

A 2015 pilot study on the Dax and Mont-de-Marsan (FERIATOX) fertilization sites on 27 patients showed that although several psychoactive substances have been identified in these patients (cocaine, ketamine, MDMA, cannabis, etc.) No DK was identified in this study. It is possible, however, that the profile of people who frequent ferias is different from that of music festivals, which explains the lack of identification of these substances in the FERIATOX study. To support this hypothesis, it seems important to renew this study on festive events of the type of music festival. The Garorock Festival (Marmande), held at the beginning of July, seems to be relevant for the study.

ELIGIBILITY:
Inclusion Criteria:

* Any patient admitted to the Emergency Medical Post with neurological and / or behavioral disorders:
* agitated at the time of admission to the PMA or during surveillance at the LDC

  * and who will say (or for whom his entourage will say that he has) consumed psychoactive substances
  * or who will be unable to say that they have taken a psychoactive substance and for which no other etiology is evident
  * and / or for which the seriousness of the case necessitates admission to the emergency or intensive care, whether or not the physician is aware of a psychoactive substance (and in the absence of an obvious etiology)
  * and / or if the PMA physician considers that analytical research is needed for further care
* Oral Express Consent
* any patient who is in possession of an identity document proving his / her majority (over 18 years).

Exclusion Criteria:

* Refusal of the patient to take a sample, or to participate in the study
* Minors (under 18 years of age)
* Pregnant women
* Breastfeeding women
* Patient who can not prove his / her age by the production of an identity document.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2017-07-03 (Actual); Study Completion 2017-07-03 (Actual)

PRIMARY OUTCOMES:
Number of patients who have consumed new psychoactive substances | baseline
  Number of patients who have consumed new psychoactive substances

SECONDARY OUTCOMES:
number of toxidomas observed clinically | Baseline
  number of toxidomas observed clinically
number of patients who have previously used new psychoactive substances (hair, urine | Baseline
  number of patients who have previously used new psychoactive substances (hair, urine
number of classes of new psychoactive substances found in the analyzes | baseline
  number of classes of new psychoactive substances found in the analyzes
severity evaluated secondarily from the clinical data sheets and according to poisoning severity score | baseline
  severity evaluated secondarily from the clinical data sheets and according to poisoning severity score

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Pellegrin, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No